CLINICAL TRIAL: NCT05892835
Title: Actitud y Conocimientos de Soporte Vital básico de Jugadores de fútbol Profesionales y Entrenadores en la Comunidad Valenciana
Brief Title: Attitude and Knowledge of Basic Life Support of Professional Soccer Players and Coaches in Valencian Community
Acronym: RCPVIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Almodóvar Fernández (Other)
Collaborators: Rafael González Moret (Unknown); Antonio Real Fernández (Unknown); Sara Simón (Unknown); Paula Sánchez Thevenet (Unknown); Hector Usó Vicent (Unknown)
Responsible Party: Sponsor-Investigator, Isabel Almodóvar Fernández, PhD, Cardenal Herrera University
Organization: Cardenal Herrera University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RCP_VIL
Record Dates: First submitted 2023-05-11; First posted 2023-06-07 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Sports Accident
Keywords: CPR; Knowledge; attitude; soccer
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: The attitude and knowledge about CPR were measured before and after the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- educative intervention (Other): A 2-hour training workshop was carried out where a theoretical explanation was given to recognize a cardiorespiratory arrest, the correct technique of chest compressions, ventilations and DESA management, in addition a practical class was carried out with CPR training models (Mannequin for CPR practices Little Anne QCPR. Laerdal) and AED simulation for CPR training (AED Practi-Trainer - Bilingual. WNL). Both theoretical and practical training were given by a basic life support instructor from the Spanish Society of Intensive Medicine and Coronary Units (SEMICYUC), the participants were instructed under the guidelines of the 2021 CKD recommendations.
  Interventions: Other: Educative

INTERVENTIONS:
Other: Educative — A 2-hour training workshop was held where a theoretical explanation was given to recognize a cardiorespiratory arrest, the correct technique of chest compressions, ventilations and DESA management, in addition a practical class was carried out with CPR training models (Manikin for CPR practices Little Anne QCPR). Laerdal and AED simulation for CPR training (AED Practi-Trainer - Bilingual. WNL). Both theoretical and practical training were given by a basic life support instructor from the Spanish Society of Intensive Medicine and Coronary Units (SEMICYUC), the participants were instructed under the guidelines of the 2021 CKD recommendations.
  Other Names: formative

SUMMARY:
Aim Given the increasing occurrence of cases of cardiorespiratory arrest on soccer fields around the world, it seems pertinent to find out the degree of training and the attitude shown by the players and coaches themselves.

The objective was to measure the knowledge and attitude of soccer professionals before and after a training intervention.

Method After an exhaustive bibliographic review, a series of questions have been analyzed and selected, with which an ad hoc questionnaire has been prepared. This questionnaire has been completed by soccer players from the Spanish first division, male and female teams and their coaches. Once the data was collected, a training workshop was carried out to improve both the attitude and knowledge in relation to cardiopulmonary resuscitation (CPR).

DETAILED DESCRIPTION:
This longitudinal descriptive study, carried out on soccer players and coaches during the year 2021. In accordance with Law 14/2007, of July 3, on biomedical research, all the data derived from this study have been treated separately from the identity of the group studied, as stated in the Declaration of Helsinki on research with human beings (2013), Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016, on natural persons in what regarding the processing of personal data and their free circulation, and Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights. The study was approved by the Ethics Committee for Biomedical Research of the CEU Cardenal Herrera University (CEEI22/286), prior approval by the medical teams of the football clubs. of the first division of the Santander League in the Valencian Community: Villarreal Club de Fútbol, Elche Club de Fútbol and Levante Unión Deportiva to participate in it. All participants gave their written consent after being informed.

After the bibliographic search of the questionnaires existing up to now to assess both the attitude of helping others and the knowledge of CPR in lay and healthcare first responders, a questionnaire was configured based on the questionnaires found due to their suitability.

After answering the questionnaire, a 2-hour training workshop was held where a theoretical explanation was given to recognize a cardiorespiratory arrest, the correct technique of chest compressions, ventilations and DESA management, in addition a practical class was carried out with CPR training models ( Manikin for CPR practices Little Anne QCPR. Laerdal) and AED simulation for CPR training (AED Practi-Trainer - Bilingual. WNL). Both theoretical and practical training were given by a basic life support instructor from the Spanish Society of Intensive Medicine and Coronary Units (SEMICYUC), the participants were instructed under the guidelines of the 2021 CKD recommendations.

One month after the training workshop, the questionnaire was passed electronically again, through a link, to obtain the post-training results.

The Shapiro-Wilk test was used to verify the normality of the variables. In case of breaking the normality condition (p<0.05) non-parametric tests were used. The calculation of each questionnaire was carried out awarding one point if the answer was correct and zero points if it was not.

ELIGIBILITY:
Inclusion Criteria: Be a professional football player or coach and agree to participate in the study -

Exclusion Criteria: Not completing the questionnaire one month after the educational intervention

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
rate the attitude in frot of CPR among the different groups | 1 month
  Rate the Knowledge and attitudes towards CPR were measured in football players and coaches.
Describe the sociodemographic parameters among the different grupos. | 1 month
  Rate and Compare the attitudes taking in acount sociodemographic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Almodóvar Fernández, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No
We are planning to send the results to "Emergencias" a Spanish journal about CPR.